CLINICAL TRIAL: NCT05106582
Title: Assessment of the Learning Curve of Total Thoracoscopic Mitral Valve Repair Using Cumulative Sum Analysis (CUSUM)
Brief Title: Assessment of the Learning Curve of Total Thoracoscopic Mitral Valve Repair
Status: Completed | Type: Observational
Sponsor: Yunlong Fan (Other)
Responsible Party: Sponsor-Investigator, Yunlong Fan, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: chinaPLAGH-08983220
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Total Thoracoscopic Mitral Valve Plasty; Minimally Invasive; Learning Curve

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total thoracoscopic mitral valve plasty (MVP) is characterized by minimal trauma, minimal bleeding, and short postoperative recovery time. The learning curve of any new procedure needs to be evaluated for learning and replication.Using Cardiopulmonary bypass (CPB) time and Aortic clamping (AC) time as evaluation variables, we visualized the learning curve for total thoracoscopic MVP using Cumulative sum analysis. We also analyzed important postoperative variables such as postoperative drainage, duration of mechanical ventilation, ICU stay and postoperative hospital stay.

The retrospective study comprised 150 consecutive patients who underwent total thoracoscopic MVP from October 2017 to July 2021.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years who underwent total thoracoscopic MVP without concurrent cardiac Surgery

Exclusion Criteria:

* data miss greater than 10%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age over 18 years who underwent total thoracoscopic MVP without concurrent cardiac Surgery
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary bypass (CPB) time | Intra-operative
  Cardiopulmonary bypass (CPB) time was used as the main variables for evaluation and visualization of the total thoracoscopic mitral valve plasty (MVP) learning curve using Cumulative sum.Cumulative sum (CUSUM) is a statistical method that focuses on results rather than on the process of performing a program skills, it generates graphs that allow for quick detection of deviations from pre-established standards and is an alternative tool that can be used to evaluate the performance of individual program. CUSUM can be generated based on set acceptable and unacceptable failure rates and the degree to which type 1(α) and type 2(β) errors (false positive and false negative errors) will be tolerated. CUSUM was defined as Sn = ∑(Xi -p0), where Xi = 0 for success and Xi = 1 for failure, p0 is the target reference.
Aortic clamping (AC) time | Intra-operative
  Aortic clamping (AC) time was used as the main variables for evaluation and visualization of the total thoracoscopic mitral valve plasty (MVP) learning curve using Cumulative sum.Cumulative sum (CUSUM) is a statistical method that focuses on results rather than on the process of performing a program skills, it generates graphs that allow for quick detection of deviations from pre-established standards and is an alternative tool that can be used to evaluate the performance of individual program. CUSUM can be generated based on set acceptable and unacceptable failure rates and the degree to which type 1(α) and type 2(β) errors (false positive and false negative errors) will be tolerated. CUSUM was defined as Sn = ∑(Xi -p0), where Xi = 0 for success and Xi = 1 for failure, p0 is the target reference.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided